CLINICAL TRIAL: NCT02245048
Title: Carotid Intima-Media Thickness and Plaque Assessment Findings in Subjects Undergoing Stress Echocardiography For Risk Stratification
Brief Title: CIMT and Plaque Assessment Findings in Subjects Undergoing Stress Echocardiography For Risk Stratification
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Esaote North America (Unknown)
Responsible Party: Principal Investigator, Tasneem Z. Naqvi, M.D., PI, Mayo Clinic
Other Study IDs: 13-008535
Record Dates: First submitted 2014-09-17; First posted 2014-09-19 (Estimated); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Cardiovascular Risk Stratification; Carotid Intima-media Thickness (CIMT); Stress Echocardiography (SE)
Keywords: Cardiovascular Risk Stratification; Carotid intima-media thickness (CIMT); Stress echocardiography (SE)
MeSH Terms: interventions — Carotid Intima-Media Thickness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stress Echocardiography (SE): Subjects will undergo CIMT measurements.
  Interventions: Other: Carotid Intima-Media Thickness (CIMT)

INTERVENTIONS:
Other: Carotid Intima-Media Thickness (CIMT)

SUMMARY:
The purpose of this research study is to determine if carotid artery ultrasound scanning can provide additional information for determining cardiovascular risk in patients.

Patients who agree to participate wil undergo non-invasive carotid intima-media thickness (CIMT) measurement and plaque assessment. Findings of CIMT will be compared to results of patient standard of care stress echocardiogram (SE) and of diastolic function.

We hypothesize tht 1) in patients undergoing SE for inappropriate or uncertain indications, CIMT and plaque assessment will provide useful risk stratification beyond use of traditional risk factors; 2) CIMT findings will correlate with results of SE in terms of exercise capacity and 3) Exercise capacity will correlate with diastolic function.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic
* No prior cardiac history (MI, PTCA, CABG, angina)
* No peripheral vascular disease
* No history of stroke or TIA
* Statins, antihypertensives, ASA treatment OK

Exclusion Criteria:

* History of CAD, CABG, PTCA, coronary or peripheral stenting
* History of stroke/TIA/peripheral vascular disease
* Inability to exercise on the treadmill
* Unwilling/unable to sign informed consent
* History of neck radiation or neck surgery or inability to obtain neck images
* End stage renal disease
* Preoperative evaluation
* History of chest pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be undergoing standard of care stress echocardiography
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
% Patients w/ Abnormal IMT vs. % Patients w/ Positive Ischemia on Stress Echocardiogram | Baseline
  We are comparing the % of patients with abnormal IMT defined as presence of plaque (= or >1.5mm) or CIMT >75% percentile for age, race, and gender compared to % of patients with positive ischemia on stress echocardiogram as defined by a new wall motion abnormality on echocardiogram with stress.

CONTACTS AND LOCATIONS:
Overall Officials: Tasneem Naqvi, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials